CLINICAL TRIAL: NCT02216240
Title: Safety and Efficacy of Paramedic Treatment of Regular Supraventricular Tachycardia
Acronym: Para-SVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: London Ambulance Service NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005795QM
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Paramedics; Standard of Care

ARMS (2):
- Accident and emergency (Active Comparator): Patients randomised to A&E were treated as per standard care and given no information other than that pertaining to the study.
  Interventions: Other: Standard care
- Paramedic (Experimental): Treatment at the scene by a paramedic. Valsalva manoeuvre with subsequent administration of 6mg and 12mg of adenosine unless the supraventricular tachycardia terminated. Patients were taken to accident and emergency if the tachycardia did not terminate, restarted, or the patient had continuing symptoms, a persistently abnormal ECG (other than T wave inversion) or was heamodynamically unstable. Prior to discharge from the ambulance patients received an information pack and a referral letter for their GP to refer them to an arrhythmia clinic.
  Interventions: Other: Paramedic

INTERVENTIONS:
Other: Paramedic
  Arms: Paramedic
Other: Standard care
  Arms: Accident and emergency

SUMMARY:
Supraventricular tachycardia (SVT) is a term describing any rhythm coming from the top half of the heart. Although atrial fibrillation is the commonest cardiac arrhythmia, regular SVT's are also common. The two commonest regular SVT's are atrioventricular (nodal) reentry tachycardias (AV(N)RT) and atrial flutter (AFL). Atrioventricular (nodal) reentry tachycardias (AV(N)RT) are common but benign forms of fast heart rhythm. Although AV(N)RT can cause unpleasant symptoms and are frightening it is not dangerous. If patients present with AV(N)RT the accepted and normal treatment for most is to have the fast heart rhythm stopped by either taking a deep breath and straining or by the use of drugs. Patients can then be discharged home and have further investigation and treatment as an outpatient. SVT can be frightening for the patient but is easy to diagnose and treat. There is high success rate post treatment for this benign condition. This is traditionally done in the local accident and emergency, although patients can sometimes be unnecessarily admitted to hospital overnight. We propose to investigate the safety and efficacy of training paramedics to treat safe forms of AV(N)RT at the scene and then giving the patient an information pack which includes a request for a GP referral to a heart rhythm specialist. Patients will be randomly allocated after consenting to take part in the study to either get paramedic or accident and emergency department treatment. We will compare these two approaches by telephone follow up of the patients. The costs of the different approaches will be compared by assessing the rate of appropriate investigation and the information given to patients and how they rated their experiences.

ELIGIBILITY:
Inclusion Patients presenting with regular narrow complex tachycardia on 12 lead ECG

Exclusion Age < 16 years Already enrolled in the study or another research study Syncope or blackout Sinus tachycardia ECG evidence of myocardial infarction Broad Complex tachycardia A history of illicit drug use within the previous 24 hours A history of structural or ischaemic heart disease Inability or unwillingness to give consent Pregnancy Failure to obtain intravenous access Hypotension - defined as a systolic blood pressure of <100 systolic Contraindications to Adenosine injection Heart transplant patients Patients on dipyridamole Patients on regular asthma inhalers Obvious atrial flutter

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-12-05 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
The cumulative time from 999 call to discharge from care for each episode of arrhythmia at 6 month follow-up | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Honarbakhsh S, Baker V, Kirkby C, Patel K, Robinson G, Antoniou S, Richmond L, Ullah W, Hunter RJ, Finlay M, Earley MJ, Whitbread M, Schilling RJ. Safety and efficacy of paramedic treatment of regular supraventricular tachycardia: a randomised controlled trial. Heart. 2017 Sep;103(18):1413-1418. doi: 10.1136/heartjnl-2016-309968. Epub 2016 Sep 9. PMID 27613170